CLINICAL TRIAL: NCT00026299
Title: A Phase I/ Randomized Phase II Trial Of Oxaliplatin (NSC #266046) With Or Without ZD 1839 (NSC # 715055) In Patients With Advanced Colorectal Carcinoma
Brief Title: Oxaliplatin With or Without Gefitinib in Treating Patients With Metastatic or Locally Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11089A; UCCRC-11089; NCI-3857
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Gefitinib; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 2: Oxaliplatin plus ZD1839 (Experimental): Oxaliplatin will be administered by IV infusion once every 21 days at a fixed dose of 130 mg/m2 and ZD1839 will be taken orally at a dose of 250 mg or 500 mg daily (as determined during phase 1). Subjects can continue to receive the combination for 6 cycles (each cycle is 21 days). After 6 cycles of the combination, subjects can continue to take ZD1839 alone until their cancer worsens.
  Interventions: Drug: ZD1839; Drug: oxaliplatin
- Phase 2: Oxaliplatin alone (Experimental): Oxaliplatin will be administered by IV infusion once every 21 days at a fixed dose of 130 mg/m2 for up to 6 cycles. Each cycle will last 21 days.
  Interventions: Drug: oxaliplatin
- Phase I: Oxaliplatin with ZD1839 (Experimental): Oxaliplatin will be administered by IV infusion once every 21 days at a fixed dose of 130 mg/m2. ZD1839 will be taken orally at a dose of 250 mg or 500 mg daily.
  Interventions: Drug: ZD1839; Drug: oxaliplatin

INTERVENTIONS:
Drug: ZD1839
  Other Names: gefitinib, Iressa ®
  Arms: Phase 2: Oxaliplatin plus ZD1839; Phase I: Oxaliplatin with ZD1839
Drug: oxaliplatin
  Other Names: Eloxatin ®

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies such as gefitinib may interfere with the growth of the tumor cells and slow the growth of colorectal cancer. Combining chemotherapy with gefitinib may kill more tumor cells.

PURPOSE: Phase I/II trial to compare the effectiveness of chemotherapy with or without gefitinib in treating patients who have metastatic or locally recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recommended phase II dose of gefitinib when administered in combination with oxaliplatin in patients with metastatic or locally recurrent colorectal cancer.
* Determine the dose-limiting toxicity of this regimen in these patients.
* Compare the time to progression, objective response rate, and median and overall survival in patients treated with oxaliplatin with or without gefitinib.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a phase I dose-escalation study of gefitinib followed by a phase II randomized, multicenter study. Patients are stratified according to ECOG performance status (0 vs 1-2).

* Phase I: Patients receive oxaliplatin IV over 2 hours on day 1 and oral gefitinib once daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gefitinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients are randomized to one of two treatment arms.

  * Arm I: Patients receive oxaliplatin IV over 2 hours on day 1.
  * Arm II: Patients receive oxaliplatin as in arm I and oral gefitinib once daily at the MTD on days 1-21.

In both arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients in arm II with stable or responding disease after 6 courses may continue to receive gefitinib alone until disease progression.

PROJECTED ACCRUAL: Approximately 77 patients (9 for phase I and 68 for phase II) will be accrued for this study within 12-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is not amenable to potentially curative surgical resection
* Metastatic or locally recurrent disease
* Tumor in liver or lung accessible to needle biopsy by ultrasound or CT scan guidance
* At least 1 measurable lesion

  * At least 20 mm by conventional techniques, including physical examination, CT scan, or MRI OR
  * At least 10 mm by spiral CT scan
  * Lesions on colonoscopic examination or barium studies, bone metastases, CNS lesions, and ascites are not considered measurable
* Failed prior therapy with fluorouracil, leucovorin calcium, and irinotecan given either sequentially or in combination
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy greater than grade 1
* No other concurrent uncontrolled illness that would preclude study
* No concurrent psychiatric illness or social situation that would preclude study
* No ongoing or active infection
* No prior allergic reaction to compounds of similar chemical or biologic composition to oxaliplatin or gefitinib
* No other concurrent malignancy except non-melanoma skin cancer or carcinoma in situ of the cervix unless considered to be at less than 30% risk of relapse after completion of therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior epidermal growth factor inhibitor
* At least 24 hours since prior colony-stimulating factors
* No concurrent colony-stimulating factors during first course of study therapy

Chemotherapy:

* See Disease Characteristics
* No more than 2 prior chemotherapy regimens for metastatic disease
* Prior adjuvant chemotherapy allowed
* At least 4 weeks since prior cytotoxic chemotherapy and recovered
* No prior cisplatin or oxaliplatin

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery

Other:

* At least 30 days since prior investigational agents
* Recovered from prior therapy
* No concurrent anti-retroviral therapy for HIV
* No other concurrent investigational or commercial agents or therapies for malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2001-09; Primary Completion 2002-12 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Recommended dose of ZD1839 in combination with oxaliplatin | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (12):
- United States (12):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan

REFERENCES:
- [Result] Kindler HL, Friberg G, Skoog L, Wade-Oliver K, Vokes EE. Phase I/II trial of gefitinib and oxaliplatin in patients with advanced colorectal cancer. Am J Clin Oncol. 2005 Aug;28(4):340-4. doi: 10.1097/01.coc.0000159558.19631.d5. PMID 16062074